CLINICAL TRIAL: NCT00275769
Title: Complete Automatic Pacing Threshold Utilization Recorded by EnPulse
Brief Title: CAPTURE - Complete Automatic Pacing Threshold Utilization Recorded by EnPulse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 229
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Arrhythmia; Bradycardia
Keywords: Arrhythmia; Bradycardia; Cardiac Pacemaker Artificial
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia

INTERVENTIONS:
Device: Pacemaker

SUMMARY:
This study compares the pacemaker's automatic pacing threshold measurements to the manual measurements conducted by a health care provider.

DETAILED DESCRIPTION:
The purpose(s) of the study is (are) to evaluate several features available in EnPulse Series pacemaker and report the long term benefit of Atrial Capture Management (ACM) and Ventricular Capture Management (VCM) as demonstrated by accuracy in comparison with manual measurements and variability of ACM and VCM thresholds.

In addition, an evaluation of the timesaving and qualitative benefits of the device feature known as Quick Look II (the computer interface screen of the device programmer) will be measured through the use of a questionnaire completed by the health care professionals involved in patient follow-up care.

This is a one-to-one randomized, multicenter, prospective study in which patients receiving new EnPulse pacemaker implants will be randomized to each of three study arms, 1) routine manual follow-up and follow-up using the automatic features; 2) ACM diagnostics detail on or VCM diagnostics detail on; 3) PMOP on / off or PMOP off / on (6 month cycle).

ELIGIBILITY:
Inclusion Criteria:

• Patients that meet ACC/AHA/NASPE 2002 class I or II dual chamber pacing indications (intended for a Pacing Mode programmed to DDD or DDDR)

Exclusion Criteria:

* Patient with mechanical tricuspid heart valves
* Patients with medical conditions that preclude the testing required by the protocol or limit study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 860
Dates: Start 2004-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The automatic device features Atrial Capture Management and Ventricular Capture Management measure pacing thresholds and is compared to manual pacing thresholds observed at the 6 month follow-up visit

SECONDARY OUTCOMES:
Observe the variability of multiple pacing thresholds measured with ACM and VCM
Observe visit time differences using automatic measurements versus traditional follow-up
Observe the effects of Post Mode Switch Overdrive Pacing (PMOP) on AT/AF burden.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen W. Mester, MD, Principal Investigator — Tampa General Hospital; Lawrence S. Rosenthal, MD, Principal Investigator — UMass Memorial Health; Raymond Gendreau, MD, Principal Investigator — Cite di la Sante de Laval
Locations (57):
- United States (51):
  - Anchorage, Alabama
  - Mobile, Alabama
  - Fullerton, California
  - Oceanside, California
  - Redondo Beach, California
  - Stanford, California
  - Colorado Springs, Colorado
  - Washington D.C., District of Columbia
  - Brandon, Florida
  - Daytona Beach, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Athens, Georgia
  - Gainsville, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Worcester, Maine
  - Burlington, Massachusetts
  - Petoskey, Michigan
  - Saint Paul, Minnesota
  - Jackson, Mississippi
  - Columbia, Missouri
  - St Louis, Missouri
  - Flemington, New Jersey
  - Newark, New Jersey
  - Paramus, New Jersey
  - Albuquerque, New Mexico
  - Fayetteville, New York
  - New York, New York
  - High Point, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Steubenville, Ohio
  - Lawton, Oklahoma
  - Tualatin, Oregon
  - Altoona, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pawtucket, Rhode Island
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Sioux Falls, South Dakota
  - Knoxville, Tennessee
  - Oak Ridge, Tennessee
  - Forth Worth, Texas
  - Houston, Texas
  - Richmond, Virginia
  - Spokane, Washington
  - Charleston, West Virginia
  - Wausau, Wisconsin
- Canada (6):
  - North Vancouver, British Columbia
  - Kitchener, Ontario
  - Toronto, Ontario
  - Laval, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Rosenthal LS, Mester S, Rakovec P, Penaranda JB, Sherman JR, Sheldon TJ, Zeng C, Wang P; CAPTURE Trial Investigators. Factors influencing pacemaker generator longevity: results from the complete automatic pacing threshold utilization recorded in the CAPTURE Trial. Pacing Clin Electrophysiol. 2010 Aug;33(8):1020-30. doi: 10.1111/j.1540-8159.2010.02809.x. Epub 2010 Jun 2. PMID 20545869